CLINICAL TRIAL: NCT05579249
Title: Effectiveness of Semaglutide 2.4 mg vs. Commercially Available Medications for Chronic Weight Management in Participants With Obesity in a Multi-employer Setting in The US - a Pragmatic Clinical Study
Brief Title: A Research Study Comparing Wegovy to Other Weight Management Drugs in People Living With Obesity in America
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9536-4741; U1111-1263-7301 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-10-11; First posted 2022-10-13 (Actual); Results first posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — semaglutide; Orlistat; Qsymia; Naltrexone; Bupropion; bupropion hydrochloride, naltrexone hydrochoride drug combination; Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Semaglutide (Experimental): Participants will receive semaglutide 2.4 milligrams (mg) subcutaneous (s.c.) injection once weekly for 52 weeks as adjuncts to a reduced-calorie diet and increased physical activity for chronic weight management.
  Interventions: Drug: Semaglutide
- Other anti-obesity medication (Active Comparator): Participants will receive one of 4 commercially available anti-obesity medication chosen by the study doctor for 52 weeks as adjuncts to a reduced-calorie diet and increased physical activity for chronic weight management. The 4 anti-obesity medications are orlistat per os [by mouth] (p.o.), phentermine/topiramate extended release p.o., naltrexone/bupropion extended release p.o. or liraglutide 3.0 mg s.c injection.
  Interventions: Drug: Orlistat; Drug: Phentermine/Topiramate; Drug: Naltrexone/Bupropion; Drug: Liraglutide

INTERVENTIONS:
Drug: Semaglutide — Participants will receive semaglutide 2.4 milligrams (mg) subcutaneous (s.c.) injection once weekly for 52 weeks.
  Other Names: Wegovy
  Arms: Semaglutide
Drug: Orlistat — Participants will receive one of 4 commercially available anti-obesity medication chosen by the study doctor for 52 weeks. The 4 anti-obesity medications are orlistat per os [by mouth] (p.o.), phentermine/topiramate extended release p.o., naltrexone/bupropion extended release p.o. or liraglutide 3.0 mg s.c injection.
  Other Names: Xenical
  Arms: Other anti-obesity medication
Drug: Phentermine/Topiramate — Participants will receive one of 4 commercially available anti-obesity medication chosen by the study doctor for 52 weeks. The 4 anti-obesity medications are orlistat per os [by mouth] (p.o.), phentermine/topiramate extended release p.o., naltrexone/bupropion extended release p.o. or liraglutide 3.0 mg s.c injection.
  Other Names: Qsymia
  Arms: Other anti-obesity medication
Drug: Naltrexone/Bupropion — Participants will receive one of 4 commercially available anti-obesity medication chosen by the study doctor for 52 weeks. The 4 anti-obesity medications are orlistat per os [by mouth] (p.o.), phentermine/topiramate extended release p.o., naltrexone/bupropion extended release p.o. or liraglutide 3.0 mg s.c injection.
  Other Names: Contrave
  Arms: Other anti-obesity medication
Drug: Liraglutide — Participants will receive one of 4 commercially available anti-obesity medication chosen by the study doctor for 52 weeks. The 4 anti-obesity medications are orlistat per os [by mouth] (p.o.), phentermine/topiramate extended release p.o., naltrexone/bupropion extended release p.o. or liraglutide 3.0 mg s.c injection.
  Other Names: Saxenda
  Arms: Other anti-obesity medication

SUMMARY:
The purpose of this post approval pragmatic clinical study is to see how well semaglutide lowers body weight compared to other medication on the market used to treat obesity, across three US-based employers. These employers represent employees of diverse demography and job functions including hospitality, clerical, administrative, housekeeping, maintenance, and specialised employees across a range of socioeconomic and educational backgrounds. The study will also look at how weight loss affects physical functioning, quality of life and ability to work. It will also gather information on how satisfied participants are with the medication they take. Participants will either receive semaglutide or one of 4 approved anti-obesity medication (Xenical/Qsymia/Contrave/Saxenda).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) greater than equal to 30.0 kilogram per meter square (kg/m^2).
* Employed at randomisation by one of the selected employers and expecting to be so for the duration of the study.

Exclusion Criteria:

* Known or suspected hypersensitivity or contraindications to Wegovy or related products according to the label.
* Known or suspected hypersensitivity or contraindications to all of the other Anti-Obesity Medications (AOMs) for chronic weight management (Xenical, Qsymia, Contrave, and Saxenda) or related products according to the labels.
* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using highly effective contraceptive method.
* History of type 1 or type 2 diabetes mellitus.
* Any disorder, unwillingness, or inability, not covered by any of the other exclusion criteria, which in the investigator's opinion might jeopardise participant's safety or compliance with protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2023-01-19 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Nutrition Research Centre, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at one site in United States.
Groups:
- Semaglutide 2.4 mg: Participants received once weekly semaglutide 2.4 milligrams (mg) subcutaneous (s.c) injection for 52 weeks as adjuncts to a reduced-calorie diet and increased physical activity for chronic weight management.
- Other Anti-obesity Medications (AOMs): Participants received one of 4 commercially available anti-obesity medication chosen by the study doctor for 52 weeks as adjuncts to a reduced-calorie diet and increased physical activity for chronic weight management. The 4 anti-obesity medications were orlistat per os [by mouth] (p.o.), phentermine/topiramate extended release p.o., naltrexone/bupropion extended release p.o. or liraglutide 3.0 mg s.c injection.
Period: Overall Study
Arm/Group | Semaglutide 2.4 mg | Other Anti-obesity Medications (AOMs)
Started | 250 | 250
Full Analysis Set | 250 | 250
Safety Analysis Set | 242 | 242
Completed | 214 | 191
Not Completed | 36 | 59
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lost to Follow-up | 33 | 52
Not completed — Physician Decision | 2 | 2
Not completed — Death | 0 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide 2.4 mg | Other Anti-obesity Medications (AOMs) | Total
Number analyzed (Participants) | 250 | 250 | 500
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.6 (9.3) | 42.0 (10.3) | 41.3 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 225 | 223 | 448
  Male | 25 | 27 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 159 | 150 | 309
  Not Hispanic or Latino | 91 | 100 | 191
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 10 | 8 | 18
  Asian | 17 | 7 | 24
  Native Hawaiian or Other Pacific Islander | 5 | 1 | 6
  Black or African American | 23 | 27 | 50
  White | 193 | 202 | 395
  More than one race | 2 | 5 | 7
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved Greater Than or Equal to (≥) 10.0 Percent (%) Body Weight Reduction (Yes/no)
Description: Number of participants who achieved greater than or equal to 10.0% body weight reduction (yes/no) at week 52 is presented.
Time Frame: At end of treatment (week 52)
Population: Full analysis set included all randomized participants. Overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Other Anti-obesity Medications (AOMs)
Number analyzed (Participants) | 207 | 177
Participants
  Yes | 132 | 61
  No | 75 | 116
Statistical Analysis 1: Comparison: Semaglutide 2.4 mg vs Other Anti-obesity Medications (AOMs); Week 52 responses were analysed using a binary regression model with randomized treatment as factor and baseline body weight as covariate; Test type: Superiority; p < 0.0001, Regression, Linear; Odds Ratio (OR) = 3.18, 95% CI 2-sided [2.12 to 4.78]

2. Secondary Outcome: Percentage Change in Body Weight
Description: Percentage change in body weight from week 0 to week 52 is presented.
Time Frame: Baseline (week 0), end of treatment (week 52)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentange change in body weight
Arm/Group | Semaglutide 2.4 mg | Other Anti-obesity Medications (AOMs)
Number analyzed (Participants) | 207 | 177
Percentange change in body weight | -13.6 (8.7) | -7.4 (7.3)

3. Secondary Outcome: Change in Impact of Weight on Quality of Life-Lite-Clinical Trials Version (IWQOL-Lite-CT) Physical Function Domain
Description: The IWQOL-Lite-CT is a 20-item, obesity-specific patient-reported outcome (PRO) instrument developed for use in obesity clinical trials. It assesses 2 primary domains of obesity-related health-related quality of life (HRQoL): physical (7 items), and psychosocial (13 items). A 5-item subset of the physical domain, the physical-function composite is also supported. Items in the physical-function composite describe physical impacts related to general and specific physical activities. All items in the physical domain are rated on either a 5-point frequency ("never" to "always") scale or a 5-point truth ("not at all true" to "completely true") scale. Total score of IWQOL-Lite-CT composite ranges from 0 to 100, with higher scores reflecting better quality of life. This outcome measure shows results for physical function domain.
Time Frame: Baseline (week 0), end of treatment (week 52)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide 2.4 mg | Other Anti-obesity Medications (AOMs)
Number analyzed (Participants) | 189 | 163
Score on a scale | 25.6 (21.2) | 22.6 (24.4)

4. Secondary Outcome: Number of Participants Who Achieved Greater Than or Equal to (≥) 15.0% Body Weight Reduction (Yes/no)
Description: Number of participants who achieved more than or equal to 15.0% body weight reduction (yes/no) at week 52 is presented.
Time Frame: At end of treatment (week 52)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Other Anti-obesity Medications (AOMs)
Number analyzed (Participants) | 207 | 177
Participants
  Yes | 93 | 25
  No | 114 | 152

5. Secondary Outcome: Number of Participants Who Achieved Greater Than or Equal to (≥) 20.0% Body Weight Reduction (Yes/no)
Description: Number of participants who achieved more than or equal to 20.0% body weight reduction (yes/no) at week 52 is presented.
Time Frame: At end of treatment (week 52)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Other Anti-obesity Medications (AOMs)
Number analyzed (Participants) | 207 | 177
Participants
  Yes | 49 | 8
  No | 158 | 169

6. Secondary Outcome: Number of Participants Who Achieved Change in Impact of Weight on Quality of Life-Lite-Clinical Trials Version (IWQOL-Lite-CT) Physical Function Domain Score Greater Than or Equal to (≥) 14.6 (Yes/no)
Description: The IWQOL-Lite-CT is a 20-item, obesity-specific patient-reported outcome (PRO) instrument developed for use in obesity clinical trials. It assesses 2 primary domains of obesity-related health-related quality of life (HRQoL): physical (7 items), and psychosocial (13 items). A 5-item subset of the physical domain, the physical-function composite is also supported. Items in the physical-function composite describe physical impacts related to general and specific physical activities. All items in the physical domain are rated on either a 5-point frequency ("never" to "always") scale or a 5-point truth ("not at all true" to "completely true") scale. Total score of IWQOL-Lite-CT composite ranges from 0 to 100, with higher scores reflecting better quality of life. This outcome measure shows results for physical function domain score ≥ 14.6.
Time Frame: At end of treatment (week 52)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Other Anti-obesity Medications (AOMs)
Number analyzed (Participants) | 189 | 163
Participants
  Yes | 138 | 108
  No | 51 | 55

7. Secondary Outcome: Percentage of Days Covered (PDC) by Study Product
Description: Percentage of days covered by study product from week 0 to week 52 is presented. The percentage of days covered by the study product is determined by the duration on the study product divided by the planned study duration, multiplied by 100.
Time Frame: From week 0 to week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of days covered
Arm/Group | Semaglutide 2.4 mg | Other Anti-obesity Medications (AOMs)
Number analyzed (Participants) | 242 | 242
Percentage of days covered | 83.7 (24.6) | 70.8 (28.6)

8. Secondary Outcome: Number of Participants Covered by Study Product Greater Than or Equal to (≥) 80% of Days (Yes/no)
Description: Number of participants covered by study product ≥80% of days (yes/no) from week 0 to week 52 is presented.
Time Frame: At end of treatment (week 52)
Population: Full analysis set included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Other Anti-obesity Medications (AOMs)
Number analyzed (Participants) | 250 | 250
Participants
  Yes | 168 | 113
  No | 82 | 137

9. Secondary Outcome: Change in Work Limitations Questionnaire 25-item Version (WLQ-25), Total Score (TS)
Description: Work Limitations Questionnaire (WLQ-25) is a 25-item questionnaire that measures how health problems affect job performance and productivity over the past two weeks, using a 5-point Likert scale. It covers four domains: Time Management (5 items), Physical Demands (6), Mental/Interpersonal (9), and Output Demands (5). Each item is scored from 1 to 5, with subscale scores calculated as the average item score, then converted to a 0-100 scale using the formula: WLQ Scale Score= 25 × (average item score - 1). Thus, each subscale ranges from 0 (no limitation) to 100 (maximum limitation). The WLQ total score is computed by applying specific weights to each subscale and summing them: 0.00048 × Time scale + 0.00036 × Physical scale + 0.00096 × Mental/Interpersonal scale + 0.00106 × Output scale. This total is then transformed into the proportion of productivity loss using the formula: (1 - exp(-total score)).
Time Frame: Baseline (week 0), end of treatment (week 52)
Population: Full analysis set included all randomized participants Overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide 2.4 mg | Other Anti-obesity Medications (AOMs)
Number analyzed (Participants) | 186 | 159
Score on a scale | -0.034 (0.070) | -0.016 (0.048)

ADVERSE EVENTS:
Time Frame: From week 0 to week 52
Description: All the presented adverse events (AEs) are treatment emergent adverse events (TEAEs). Treatment emergent adverse events (TEAEs): events that had onset date during on-treatment period, time period in which participants was considered exposed to trial product. Safety analysis set included all participants who are exposed to study intervention. AEs were assessed in SAS and All-Cause Mortality was assessed for all enrolled participants.
Arm/Group | Semaglutide 2.4 mg | Other Anti-obesity Medications (AOMs)
All-Cause Mortality (participants affected / at risk) | 0/250 | 2/250
Serious Adverse Events (participants affected / at risk) | 3/242 | 8/242
Other Adverse Events (participants affected / at risk) | 0/242 | 0/242
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 2.4 mg (N=242) | Other Anti-obesity Medications (AOMs) (N=242)
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2022-09-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT05579249/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-17): https://cdn.clinicaltrials.gov/large-docs/49/NCT05579249/SAP_001.pdf